CLINICAL TRIAL: NCT06919367
Title: Evaluation of Dental Ages of Children With Type I Diabetes Using Different Dental Age Estimation Methods-A Retrospective Cohort Study
Brief Title: Use of Dental Age Determination Methods in Children With Type Diabetes
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Deniz Sila ÖZDEMİR CELİK, Assistant Professor, Abant Izzet Baysal University
Other Study IDs: 2023/435
Record Dates: First submitted 2025-03-26; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: age estimation using orthopantomography — Dental age estimation will be performed with 3 different methods based on orthopantomographic images obtained during routine examinations of patients.

SUMMARY:
The aim of this study was to determine the estimated dental age of children with type 1 diabetes by using Cameriere, Willems and Demirjian methods.

DETAILED DESCRIPTION:
The different metabolic activities of children with type 1 diabetes cause significant differences between them and healthy children. Especially from a forensic point of view, special methods defined for these children are needed and dental age estimation is one of them. The aim of this study was to determine the estimated dental age of children with type 1 diabetes by using Cameriere, Willems and Demirjian methods.

Methods: Between 2017 and 2024, 58 patients with type 1 diabetes and healthy children were included in the study. Dental ages were calculated on panoramic radiographic images by 2 different dentists using Cameriere, Willems and Demirjian methods. Dental ages and their differences with chronological ages were compared by group and gender. Analyses were performed in IBM SPSS 25 program.

ELIGIBILITY:
Inclusion Criteria:

* 4-15 years old
* No chronic disease in addition to the diagnosis of type 1 diabetes
* Children with controlled type 1 diabetes mellitus
* No congenital tooth deficiency
* Pediatric patients with good quality panoramic radiographs were included.

Exclusion Criteria:

* Blurred or distorted radiographs,
* Missing any of the left seven permanent mandibular teeth (genesis or extraction),
* With dental abnormalities (dilaceration, supernumerary teeth) and developmental disorders (cleft lip and palate),
* Patients with incomplete medical or dental history were excluded.

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Type 1 diabetes mellitus who applied to Bolu Abant İzzet Baysal University Faculty of Dentistry Pedodontics Clinic between 2017 and 2024 were included.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2023-12-25 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
dental age estimation | 3 months
  Are the dental age prediction results of children with diabetes different from healthy children?

SECONDARY OUTCOMES:
type 1 diabetes and dental age estimation | 3 months
  What is the ideal dental age estimation method for children with type 1 diabetes?

CONTACTS AND LOCATIONS:
Locations (1):
- Abant Izzet Baysal University, Bolu, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data obtained from tooth age determination methods will be shared.